CLINICAL TRIAL: NCT02131792
Title: Early Results of Slanted Recession of the Lateral Rectus Muscle for Intermittent Exotropia With Convergence Weakness; A Prospective Study
Brief Title: Early Results of Slanted Recession of the Lateral Rectus Muscle for Intermittent Exotropia With Convergence Weakness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kyungpook National University Hospital (Other)
Responsible Party: Principal Investigator, Bo Young Chun, Department of Ophthalmology, School of medicine, Kyungpook National University, Kyungpook National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KNUH2014-02
Record Dates: First submitted 2014-05-04; First posted 2014-05-06 (Estimated); Last update posted 2014-05-06 (Estimated); Status verified 2014-05

CONDITIONS: Intermittent Exotropia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lateral Rectus Muscle Slanted Recession (Experimental): Slanted recession of the lateral rectus muscle for the intermittent exotropia with convergence weakness
  Interventions: Procedure: Slanted recession of the lateral rectus muscle

INTERVENTIONS:
Procedure: Slanted recession of the lateral rectus muscle — All patients who had intermittent exotropia with convergence weakness was enrolled to the slanted lateral rectus muscle recession group.

SUMMARY:
This study was conducted to evaluate results of slanted recession of the lateral rectus muscle for intermittent exotropia with convergence weakness

DETAILED DESCRIPTION:
This prospective study included 31 patients who underwent slanted lateral rectus muscle recession for intermittent exotropia with convergence weakness. Measurements of preoperative and postoperative deviation angle, stereopsis was performed.

ELIGIBILITY:
Inclusion Criteria:

* Patients with intermittent exotropia greater at near than at distance by 10 prism diopters or more
* Patients with follow up duration greater than 6 months

Exclusion Criteria:

* Patients with previous ocular or strabismus surgery
* Patients with ocular or neurologic pathologic conditions
* Follow up duration less than 6 months

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 31 (Actual)
Dates: Start 2010-06; Primary Completion 2012-06 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Changes from baseline of exodeviations angle after slanted recession surgery at 6 months. | preop, 6months postop
  Measurement of deviation angle after slanted recession surgery was performed.

SECONDARY OUTCOMES:
Changes from baseline of near-distance difference after slanted recession surgery at 6 months | preop, 6 months postop
  Measurement of stereopsis after slanted recession was performed.

CONTACTS AND LOCATIONS:
Overall Officials: Bo Young Chun, M.D, Principal Investigator — Kyungpook National University Hospital
Locations (1):
- Bo Young Chun, Daegu, Kyungsangpookdo, South Korea